CLINICAL TRIAL: NCT03615807
Title: Randomized Study Comparing Different Durations of Antibiotic Treatment for Diabetic Foot Infections
Brief Title: Less Infections for the Diabetic Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Ilker Uckay, Prof. Dr. med Ilker Uçkay, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: n° 2016-01008
Record Dates: First submitted 2017-01-16; First posted 2018-08-06 (Actual); Results first posted 2020-06-01 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Diabetic Foot
Keywords: diabetic foot infections; antibiotic reduction; osteomyelitis; soft tissue infections
MeSH Terms: conditions — Diabetic Foot; Osteomyelitis; Soft Tissue Infections

STUDY DESIGN:
Intervention Model Description: Two prospected-randomized protocols
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short antibiotic arm (Experimental): 10 days for soft tissue infections 3 weeks for osteomyelitis
  Interventions: Procedure: Surgical debridement (if needed); Diagnostic Test: Microbiological sampling; Procedure: Revascularisation (if needed).; Device: Off-loading; Behavioral: Patient's education and instructions; Procedure: Wound debridement; Drug: Antibiotic duration
- Standard antibiotic arm (Active Comparator): 20 days for soft tissue infections 6 weeks for osteomyelitis
  Interventions: Procedure: Surgical debridement (if needed); Diagnostic Test: Microbiological sampling; Procedure: Revascularisation (if needed).; Device: Off-loading; Behavioral: Patient's education and instructions; Procedure: Wound debridement; Drug: Antibiotic duration

INTERVENTIONS:
Procedure: Surgical debridement (if needed) — Surgical debridement
Diagnostic Test: Microbiological sampling — Microbiological sampling
Procedure: Revascularisation (if needed). — Revascularisation (if needed).
Device: Off-loading — Off-loading by Special shoes
Behavioral: Patient's education and instructions — Patient's education and instructions by specialized nurses
Procedure: Wound debridement — Regular wound debridement by specialized nurses
Drug: Antibiotic duration — Systemic antibiotic duration according to the study arms

SUMMARY:
This is a randomized, unblinded, single-centre study. After eventual surgical debridement (not amputation), patients will be randomized to receive 1 of 2 targeted antibiotic regimens, in the ratio 1:1.

For diabetic toe osteomyelitis, the patients will be randomized between a 3 and a 6 week's arm, for soft tissue infections between 10 and 20 days. The final assessments used in the primary efficacy analysis will be obtained at the test-of-cure (TOC) visit approximately 60 days after treatment is stopped.

DETAILED DESCRIPTION:
Diabetic foot infections (DFI) are frequent and are associated with a high burden of morbidity, costs, recurrence risk or new episodes of infections. About two-third of recurrent DFI may reveal other microorganisms than in the previous period, suggesting new episodes of infection due to the underlying problem, and/or selection by prior antimicrobial therapy. Osteomyelitis in the diabetic toe is almost always established by contiguous spread of infection from a chronic ulcer. It occurs in up to 15% of patients with a diabetic foot ulcer and about 20% of all DFI (and over half of severe infections) involve bone at presentation. The severity of a diabetic foot infection is based on the local and systemic signs and symptoms of infection and has been categorically defined in the Infectious Disease Society of America guidelines for the "Diagnosis and Treatment of Diabetic Foot Infections" (IDSA guidelines).

Knowing the potential for poor outcomes, many clinicians have tended to treat DFIs with a long duration of antibiotic therapy, with many side effects, development and spreading of antibiotic resistance, and associated costs. Data from recent comparative trials has shown that 1-2 weeks is sufficient for most soft tissue infections, and 4 to 6 weeks appears adequate in those with (unresected) infected bone. Retrospective reviews over the past two decades have demonstrated that about two-thirds of selected patients with diabetic foot osteomyelitis can achieve remission with antibiotic therapy alone (i.e., without bone resection). One recent randomized trial found that treatment with only antibiotic therapy (given for 90 days) gave similar clinical outcomes to treatment with conservative surgery (removal only of the infected bone) along with just a short course of antibiotic therapy. Another randomized trial compared a 6-week against 12-week course of antibiotic therapy, without concomitant surgery, for diabetic foot osteomyelitis and also found similar outcomes.

Likewise, the optimal antibiotic duration for any skin and soft tissue infection is unknown. According to some databases of University of Geneva Hospitals, among 378 skin and soft tissue infections in 346, overall cure was achieved in 330 episodes (87%) after a median antibiotic administration of 15 days. In multivariate Cox regression analysis, duration of antibiotic therapy (HR 1.0, 95%CI 0.96-1.02) did not influence treatment failure among patients with positive MRSA carriage.

Our study intends to optimize the duration of antibiotic therapy in DFI; for skin and soft tissue infections as well as for diabetic toe osteomyelitis that is not amputated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Diabetes mellitus
3. Diabetic Foot Infections
4. Surgical intervention to remove all necrotic tissue or tenotomy.
5. Osteomyelitis limited to bone contact or cortical lesions in X-ray.

Exclusion Criteria:

1. Implanted device.
2. More than 96 hours of systemic antibiotic therapy prior to inclusion
3. Amputation
4. Destructive osteomyelitis
5. Concomitant infections requiring more than 14 days of antibiotic therapy.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Uçkay, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tone A, Nguyen S, Devemy F, Topolinski H, Valette M, Cazaubiel M, Fayard A, Beltrand E, Lemaire C, Senneville E. Six-week versus twelve-week antibiotic therapy for nonsurgically treated diabetic foot osteomyelitis: a multicenter open-label controlled randomized study. Diabetes Care 2015;38:302-307. Diabetes Care. 2015 Apr;38(4):735. doi: 10.2337/dc15-er04b. No abstract available. PMID 25805867
- [Derived] Pham TT, Gariani K, Richard JC, Kressmann B, Jornayvaz FR, Philippe J, Lipsky BA, Uckay I. Moderate to Severe Soft Tissue Diabetic Foot Infections: A Randomized, Controlled, Pilot Trial of Post-debridement Antibiotic Treatment for 10 versus 20 days. Ann Surg. 2022 Aug 1;276(2):233-238. doi: 10.1097/SLA.0000000000005205. Epub 2021 Sep 15. PMID 35623048
- [Derived] Gariani K, Pham TT, Kressmann B, Jornayvaz FR, Gastaldi G, Stafylakis D, Philippe J, Lipsky BA, Uckay L. Three Weeks Versus Six Weeks of Antibiotic Therapy for Diabetic Foot Osteomyelitis: A Prospective, Randomized, Noninferiority Pilot Trial. Clin Infect Dis. 2021 Oct 5;73(7):e1539-e1545. doi: 10.1093/cid/ciaa1758. PMID 33242083

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Short Antibiotic Arm | Standard Antibiotic Arm
Started | 91 | 91
Completed | 79 | 80
Not Completed | 12 | 11

BASELINE CHARACTERISTICS:
Population: Diabetic foot infections requiring tretement
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Antibiotic Arm | Standard Antibiotic Arm | Total
Number analyzed (Participants) | 79 | 80 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 38 | 65
  >=65 years | 52 | 42 | 94
Age, Continuous [Median (Full Range); unit: years] | 70 [38 to 90] | 67 [34 to 94] | 68 [34 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 70 | 72 | 142
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 79 | 80 | 159
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 79 | 80 | 159

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Clinical Failure
Description: Visual and dichotomous evaluation regarding the numbers of clinical recurrence/failure
Time Frame: 30-60 days
Measure: Number; unit: Participants
Groups:
- Short Antibiotic Arm: For soft tissue infection: 10 days of systemic antibiotics For osteomyelitis: 3 weeks
- Long Antibiotic Arm: For soft tissue infections: 20 days For osteomyelitis: 6 weeks
Arm/Group | Short Antibiotic Arm | Long Antibiotic Arm
Number analyzed (Participants) | 79 | 80
Participants | 26 | 30

2. Secondary Outcome: Number of Participants Experiencing Adverse Events Related to the Antibiotic Therapy
Description: Adverse events related to the antibiotic therapy.
Time Frame: 30-60 days
Measure: Number; unit: Participants
Arm/Group | Short Antibiotic Arm | Long Antibiotic Arm
Number analyzed (Participants) | 79 | 80
Participants | 31 | 27

ADVERSE EVENTS:
Time Frame: The adverse events were collected during the first two months of therapy.
Description: Adverse Events Definition: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Short Antibiotic Arm: 10 days antibiotic for soft tissue infections 3 weeks antibiotic for osteomyelitis
- Long Antibiotic Arm: 20 days antibiotic for soft tissue infections 6 weeks antibiotic for osteomyelitis
Arm/Group | Short Antibiotic Arm | Long Antibiotic Arm
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/80
Serious Adverse Events (participants affected / at risk) | 5/79 | 6/80
Other Adverse Events (participants affected / at risk) | 5/79 | 6/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Antibiotic Arm (N=79) | Long Antibiotic Arm (N=80)
Progressive ischemia leading to necrosis and amputation (General disorders) | 5 (5) | 6 (6) — Progressive ischemia leading to necrosis and amputation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Antibiotic Arm (N=79) | Long Antibiotic Arm (N=80)
Cutaneous rash (General disorders) | 5 (5) | 6 (6) — Cutaneous rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT03615807/Prot_SAP_000.pdf